CLINICAL TRIAL: NCT05758857
Title: Multiple Risk Factor Intervention Trial: A Pilot Study
Brief Title: Multiple Risk Factor Intervention Trial
Acronym: Ms FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Amy Kirkham, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 43521
Record Dates: First submitted 2023-02-03; First posted 2023-03-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Metabolic Disturbance; Sedentary Behavior
Keywords: primary prevention
MeSH Terms: conditions — Sedentary Behavior | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: 3-arm parallel-group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind participants to their assigned intervention. Care providers are not involved. The outcome assessors for any assessments involving potential for subjectivity in data collection or analysis will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guidelines-based physical activity (Experimental): 150 weekly minutes of moderate-intensity aerobic activity and twice weekly whole-body muscle strengthening
  Interventions: Behavioral: Experimental: Guidelines-based physical activity
- Guidelines-based physical activity and healthy eating (Experimental): 150 weekly minutes of moderate-intensity aerobic activity and twice weekly whole-body muscle strengthening + counselling to follow Canada's Food Guide
  Interventions: Behavioral: Experimental: Guidelines-based physical activity; Behavioral: Experimental: Guidelines-based healthy eating
- Stretching exercise (Placebo Comparator): Whole-body stretching
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Experimental: Guidelines-based physical activity — Through a combination of exercise trainer-led in-person and virtual sessions, as well as counselling for independent aerobic exercise, participants will be guided to achieve 150 weekly minutes of moderate-intensity aerobic activity and twice weekly whole-body muscle strengthening.
  Arms: Guidelines-based physical activity; Guidelines-based physical activity and healthy eating
Behavioral: Experimental: Guidelines-based healthy eating — One-on-one phone/virtual counselling from a registered dietitian to change dietary habits to be in line with Canada's Food Guide.
  Arms: Guidelines-based physical activity and healthy eating
Behavioral: Stretching exercise — Twice weekly virtual instructor-led whole-body stretching class.
  Arms: Stretching exercise

SUMMARY:
Ms. FIT pilot is a pilot study of a 3-arm RCT with equal recruitment and stratification of pre and postmenopausal women with risk factors for chronic disease to: 1) Canadian guidelines-based physical activity alone; 2) Canadian guidelines-based physical activity and healthy eating; or 3) stretching attention control. The purpose of this study is to evaluate the feasibility, acceptability, and preliminary efficacy of the interventions. The objectives are to: 1) pilot test the intervention delivery protocol in a real-world application (management and technical capabilities of the research group); 2) evaluate adherence and participant acceptability of a combined in-person and virtual intervention delivery in both pre and post-menopausal women; 3) identify the preliminary efficacy of the interventions on select cardiometabolic risk markers.

ELIGIBILITY:
Inclusion Criteria:

* females
* pre- or postmenopausal
* aged 30+ years
* moderate or high Canadian Diabetes Risk Score score

Exclusion Criteria:

* diagnoses of cardiovascular diseases, type 2 diabetes, non-alcoholic fatty liver disease, cancer (except for non-melanoma skin cancer), or respiratory disease (i.e., COPD)
* major signs or symptoms (regardless of known diagnosis) of cardiovascular diseases, diabetes, or renal disease
* pregnant or lactating
* mobility limitations to exercise
* smoking cigarettes within the past 3 months
* using transdermal hormones, taking exogenous hormones or receiving exogenous hormones from other means (e.g. intrauterine device)
* self-report of >30 min/week of MVPA
* following a specific dietary practice (e.g., vegan, ketogenic) in last 3 months
* presenting with any of the American Heart Association's absolute or relative contraindications for symptom-limited maximal exercise testing
* requiring and do not receive medical clearance for maximal exercise
* cannot read and understand the consent form or communicate in English
* individuals who are students in classes of the professors who are involved in the study or students with whom the professors have a supervisory relationship

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Physical activity intervention feasibility | end of week 6
  Determined as an average adherence to physical activity guidelines of ≥100% measured via Garmin smartwatch
Diet quality intervention feasibility | end of week 6
  Determined as a 5-point improvement in diet quality measured via healthy eating index from 3-day diet record
Intervention acceptability | end of week 6
  Assessed via researcher-developed questionnaire

SECONDARY OUTCOMES:
Systemic insulin resistance | 6 weeks
  As assessed by the Matsuda Index calculated from an oral glucose tolerance test
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 6 weeks
  calculated as: (fasting insulin*fasting glucose)/22.5
Framingham 10-year risk (%) | 6 weeks
  Calculated using standardized scoring system
Lipid profile | 6 weeks
  analyzed from blood
C-Reactive Protein | 6 weeks
  analyzed from blood
Blood pressure | 6 weeks
  Measured after several minutes of supine rest
Aortic stiffness (central to femoral) | 6 weeks
  Measured via Shygmacor device
Brachial artery endothelial function | 6 weeks
  Measured via flow-mediated dilatation test
Cardiorespiratory fitness | 6 weeks
  Measured as peak volume of oxygen consumption via indirect calorimetry
Whole-body fat and fat free mass | 6 weeks
  Measured by BodPod
Body circumferences | 6 weeks
  Waist, hip and neck circumferences measured by inelastic tape
Depressive symptoms | 6 weeks
  measured by Beck Depression Inventory; score ranges from 0-63 with a higher score indicating more severe depression
Dietary intake | 6 weeks
  Assessed via ASA-24 3-day food records
Menopausal symptom presence and severity | 6 weeks
  assessed by The Menopause-specific Quality of Life (MENQOL) questionnaire. Each of four domains is constrained between 1 to 8 where a higher score indicates more symptoms.
Health-related quality of life | 6 weeks
  Assessed by RAND-36, where an independent score is provided for 8 scales ranging from 0 to 100 with a higher score indicating better quality of life
Psychosocial stress | 6 weeks
  assessed by the perceived stress scale where individual scores can range from 0 to 40 with higher scores indicating higher perceived stress

OTHER OUTCOMES:
Health-related quality of life | 6 months
  Assessed by RAND-36, where an independent score is provided for 8 scales ranging from 0 to 100 with a higher score indicating better quality of life
Psychosocial stress | 6 months
  assessed by the perceived stress scale where individual scores can range from 0 to 40 with higher scores indicating higher perceived stress
Intervention acceptability | 6 months
  Assessed via researcher-developed questionnaire
Menopausal symptom presence and severity | 6 months
  assessed by The Menopause-specific Quality of Life (MENQOL) questionnaire. Each of four domains is constrained between 1 to 8 where a higher score indicates more symptoms.
Dietary intake | 6 months
  Assessed via ASA-24 3-day food records
Depressive symptoms | 6 months
  measured by Beck Depression Inventory; score ranges from 0-63 with a higher score indicating more severe depression
Body circumferences | 6 months
  Waist, hip and neck circumferences measured by inelastic tape
Whole-body fat and fat free mass | 6 months
  Measured by BodPod
Cardiorespiratory fitness | 6 months
  Measured as peak volume of oxygen consumption via indirect calorimetry
Blood pressure | 6 months
  Measured after several minutes of supine rest
Physical activity intervention feasibility | 6 months
  Determined as an average adherence to physical activity guidelines of ≥100% measured via Garmin smartwatch
Diet quality intervention feasibility | 6 months
  Determined as a 5-point improvement in diet quality measured via healthy eating index from 3-day diet record

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No